CLINICAL TRIAL: NCT07165093
Title: Diagnostic Yield of Cardiac CT to Detect Cardiac Thrombi in Acute Ischemic Stroke: an Individual Patient Data Meta-Analysis
Acronym: AIS of HEARTS
Status: Completed | Type: Observational
Sponsor: Academisch Medisch Centrum - Universiteit van Amsterdam (AMC-UvA) (Other)
Responsible Party: Principal Investigator, Jonathan Coutinho, Principal Investigator, Academisch Medisch Centrum - Universiteit van Amsterdam (AMC-UvA)
Other Study IDs: NL64139.018.18
Record Dates: First submitted 2025-08-09; First posted 2025-09-10 (Actual); Last update posted 2026-01-21 (Actual); Status verified 2025-08

CONDITIONS: Ischemic Stroke; Cardioembolic Stroke; Thrombus; Cardiac CT
Keywords: cardiac CT; ischemic stroke; cardioembolic stroke; cardioembolic sources; cardiac thrombus; imaging
MeSH Terms: conditions — Ischemic Stroke; Embolic Stroke; Thrombosis

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Other
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (4):
- Amsterdam UMC: Patients from Amsterdam UMC that underwent ECG-gated cardiac CT
- Christchurch Hospital: Patients from Christchurch hospital that underwent non-ECG gated cardiac CT
- John Hunter Hospital: Patients from John Hunter Hospital that underwent non-ECG gated cardiac CT
- Liverpool Hospital: Patients from Liverpool Hospital that underwent ECG-gated cardiac CT

SUMMARY:
The aim of the AIS of HEARTS registry is to establish a database to collect, maintain and provide accessible individual patient data from international cohorts and to provide pooled analyses about the yield and value of cardiac computed tomography (CT), acquired during the initial stroke imaging protocol.

The main analysis will investigate the diagnostic yield of cardiac CT to detect cardioembolic sources of stroke in acute ischemic stroke patients.

DETAILED DESCRIPTION:
This study is an individual patient data meta-analysis of four different cohorts (4 hospitals) with both prospective and retrospective data. Patients are included if they underwent cardiac CT (ECG gated or non-ECG gated) acquired during the acute stroke scan protocol. The main paper will focus on the diagnostic yield of cardiac thrombi detected on cardiac CT acquired during the acute stroke scan protocol, the comparison with echocardiography and the 90 day follow-up outcomes.

Prospectively planned subanalyses from the AIS of HEARTS registry:

Beyond the analyses focussed on cardiac thrombi, the investigators have prespecified the following analyses:

* Risk stratification of cardioembolic sources in acute ischemic stroke to improve decision making in performing a cardiac CT
* Short term clinical implications of cardiac thrombi detected on cardiac CT
* Long term clinical implications of cardiac thrombi detected on cardiac CT
* Diagnostic yield of ECG-gated versus non-ECG-gated cardiac CT in the acute phase of ischemic stroke
* Association between left atrial appendage contrast filling characteristics and recurrent stroke
* Association between left atrial appendage (LAA) morphology/volume and LAA thrombus
* Cardiac thrombus and associations with medium vessel occlusions strokes
* High-risk cardioembolic sources on cardiac CT in TIA patients
* Clinical relevance of valvular vegetations detected on cardiac CT
* Long term clinical implications of left atrial diverticula detected on cardiac CT
* Incidental findings on cardiac CT The investigators are planning to perform these additional analyses once the main paper has been accepted/submitted.

ELIGIBILITY:
Inclusion Criteria:

* Age 18 years or older
* Clinical diagnosis of acute ischemic stroke
* Cardiac CT acquired during acute stroke scan protocol

Exclusion Criteria:

* Transient ischemic attack
* Stroke mimics

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients 18 years or older with acute ischemic stroke that underwent a cardiac CT during the acute stroke scanprotocol.
Sampling Method: Non-Probability Sample
Enrollment: 3940 (Actual)
Dates: Start 2018-05-19 (Actual); Primary Completion 2024-06-30 (Actual); Study Completion 2025-09-01 (Actual)

PRIMARY OUTCOMES:
Proportion of patients with cardiac thrombus detected on acute cardiac CT. | Baseline: the assessment of a cardiac thrombus is performed when the patient arrives at the Emergency Department and undergoes the acute stroke imaging protocol including a cardiac CT.
  The proportion of patients with acute ischemic stroke that have a cardiac thrombus detected on cardiac CT.

SECONDARY OUTCOMES:
Comparison between cardiac CT and echocardiography for the detection of cardiac thrombi. | An average of within 1 year: the investigators include echocardiography that is performed in routine stroke clinical care. This means that the time delay is dependent on various aspect of the local center.
  Proportion of acute ischemic stroke patients with a cardiac thrombus on cardiac CT and echocardiography, in patients that underwent both investigations.
Follow up 90 days: mortality compared between patients with and without thrombus | From stroke onset until 90 days follow-up
  Proportion of patients that died at 90 days follow-up after stroke onset.
Follow-up 90 days: recurrent stroke | Stroke onset until 90 days follow-up
  Proportion of patients that had a recurrent stroke at 90 days follow-up after stroke onset. A recurrent stroke needs to be clearly defined, based on clinical, imaging and other diagnostic information
Follow-up 90 days: outcome using modified rankin scale score | Stroke onset until 90 days follow-up
  Functional outcome at 90 days, measured using the modified rankin scale (mRS) score. The mRS score is a scale from 0-6. Higher scores mean a worse functional outcome.

CONTACTS AND LOCATIONS:
Overall Officials: Jonathan Coutinho, MD, PhD, Principal Investigator — Amsterdam UMC
Locations (1):
- Amsterdam UMC, Amsterdam, Netherlands

IPD SHARING:
Plan to Share IPD: Undecided